CLINICAL TRIAL: NCT01578109
Title: A Pilot Study of Sorafenib in Patients With Acute Myeloid Leukemia as Peri-Transplant Remission Maintenance
Brief Title: Sorafenib Tosylate Before and After Donor Bone Marrow Transplant in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00727; NCI-2012-00727 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J11116; CDR0000730684; 8992 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8992 (Other: CTEP); P01CA015396 (NIH); P30CA006973 (NIH); P50CA100632 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation
MeSH Terms: interventions — Bone Marrow Transplantation; Blood Specimen Collection; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sorafenib tosylate and transplant) (Experimental): Patients receive sorafenib tosylate PO BID beginning at least 30 days after completion of induction therapy and/or transplant and no more than 120 days after transplant continuing for up to 2 years after transplant in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Bone Marrow Transplantation; Drug: Sorafenib; Drug: Sorafenib Tosylate

INTERVENTIONS:
Procedure: Bone Marrow Transplantation — Undergo BMT
  Other Names: Blood and Bone Marrow Transplant; BMT; Bone Marrow Grafting; Bone Marrow Transplant; Marrow Transplantation
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43-9006; Bay-439006
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This pilot clinical trial studies the side effects of sorafenib tosylate before and after donor bone marrow transplantation in treating patients with acute myeloid leukemia. Sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the toxicity and safety of incorporation of sorafenib tosylate (sorafenib) into the pre- or post-transplant maintenance setting for three types of transplants.

SECONDARY OBJECTIVES:

I. Improvement of 2 year disease free survival after bone marrow transplant by 25% based on a baseline relapse free survival at two years of 30%.

II. Secondary graft failure is defined as the decline in neutrophil count to < 500/cu mm after achieving engraftment which is unrelated to infection or drug effect (sorafenib?) and is unresponsive to stimulation by growth factors.

III. Non-relapse mortality (NRM) is defined, as death in the absence of competing risks, relapse or progression of disease.

IV. Survival without relapse or death (disease-free survival [DFS]) or without death (overall survival [OS]) will be determined and presented as Kaplan-Meier estimates at 1 and 2 years post-transplant.

V. Patients will be evaluated for chronic graft versus host disease (GVHD) both as described in the National Institutes of Health (NIH) consensus project guidelines and by conventional criteria.

LABORATORY CORRELATIVE OBJECTIVE:

I. Patients will undergo serial examinations of bone marrow during the maintenance treatments evaluating minimal residual disease (MRD) by flow cytometry and FLT3 suppression by western blot analysis and plasma inhibitory assay (PIA).

OUTLINE: This is a dose-escalation study.

Patients receive sorafenib tosylate orally (PO) twice daily (BID) beginning at least 30 days after completion of induction therapy and/or transplant but no more than 120 days after transplant continuing for up to 2 years after transplant in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia with a FLT3-internal tandem duplication (ITD) who are in a complete remission or partial remission (less than 10% blasts in marrow) as documented by bone marrow biopsy and who plan to undergo a bone marrow transplantation
* Patients who have had count recovery (absolute neutrophil count [ANC] > 500,000/mm^3; non transfused platelet count over 30,000/mm^3) and are at least 30 days after induction and/or transplantation but no more than 120 days post transplant
* Patients may have received any prior therapy deemed necessary for induction of remission except for patients whom have progressed while on sorafenib; patients who have responded to sorafenib previously are eligible for enrollment on the protocol
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than four months
* Total bilirubin less than 2 x upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional upper limit of normal
* Creatinine =< 1.5 x upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x upper limit of normal
* The effects of sorafenib on the developing human fetus are unknown; for this reason and because tyrosine kinase inhibiting agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; contraception should continue for at least 30 days after the last dose of sorafenib
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks except for intrathecal chemotherapy (i.e., methotrexate, cytarabine, or thiotepa)
* Patients may not be receiving any other investigational agents
* Patients with uncontrolled hypertension (i.e., persistent grade 3 while undergoing treatment)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* Patients with active and/or untreated central nervous system (CNS) leukemia will not be eligible
* Patients must not have any evidence of bleeding diathesis or be on any therapeutic anticoagulation such as low molecular weight (LMW) heparin or warfarin for deep vein thrombosis (DVT) treatment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because sorafenib is chemotherapeutic agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sorafenib, breastfeeding should be discontinued if the mother is treated sorafenib
* Human immunodeficiency virus (HIV)-positive patients are excluded because management of these patients in the hematopoietic cell transplant setting has not yet been well defined and is currently the subject of investigation in other studies addressing this issue
* Patients with active acute GVHD who have been initiated on therapy or had therapy escalation within 21 days are not eligible
* Patients with lack of engraftment (less than 90% donor deoxyribonucleic acid [DNA] in bone marrow or peripheral blood) after bone marrow transplant as evidence by RFLP (restriction fragment length polymorphism) are not eligible
* Patients who are unable to swallow pills are not eligible
* Patients taking strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors including enzyme-inducing anti-epileptic drugs (phenytoin, carbamazepine, or phenobarbital), rifampin, grape fruit juice, or St. John's wort are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients removed from the study in each cohort due to toxicity | Up to 24 months
  Will be reported with exact binomial proportions and 95% confidence intervals. All toxicities by type and grade will be reported. The proportion of patients with graft failure in each cohort will also be reported with exact binomial proportions and 95% confidence intervals.

SECONDARY OUTCOMES:
Cumulative incidence of non-relapse mortality and relapse | Up to 2 years
  Estimated by competing risks analysis using Grey's method.
Disease-free survival (DFS) | Up to 2 years
  Standard life table methods with Kaplan-Meier (KM) plots will be used to analyze DFS. Reported with 90% confidence intervals overall and by cohort.
Overall survival (OS) | Up to 2 years
  Standard life table methods with KM plots will be used to analyze OS. Reported with 90% confidence intervals overall and by cohort.
Change in minimal residual disease (MRD) | Baseline to day 365
  Will be assessed by flow cytometry. Box plots will be used.
Change in FLT3 suppression | Baseline to day 365
  Will be assessed by plasma inhibitory assay and western blotting. Box plots will be used.
Pharmacodynamic parameters of sorafenib tosylate | Up to 2 years post-transplant
  Samples will be collected to assess sorafenib tosylate and the N-oxide metabolite (total and unbound) exposure to correlate with pharmacodynamic endpoints using non-parametric statistics.

OTHER OUTCOMES:
Changes in T-regulatory cell population | Baseline to 2 years post-transplant
  Regression modeling of subdistribution functions in competing risks by Gray's method will be conducted to examine how changes in immunologic parameters are associated with subsequent development of acute graft versus host disease. An appropriate transformation will be used to normalize the data. Differences between pre- and post-transplantation will be explored using methods appropriate for paired data. Patterns of change in marker values over time may also be explored using appropriate modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lewis, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (2):
- United States (2):
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland